CLINICAL TRIAL: NCT01951144
Title: A Double Blind (3rd Party Open) Randomized, Placebo Controlled, Crossover Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PF-06372865 in Healthy Male and Female Subjects
Brief Title: A First In Human Study In Healthy People To Evaluate Safety, Toleration, Pharmacokinetics and Pharmacodynamics of Single Oral Doses Of PF-06372865
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B7431001
Record Dates: First submitted 2013-09-13; First posted 2013-09-26 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Phase 1; Single Dose; Pharmacokinetics; Safety; Toleration; Pharmacodynamics
MeSH Terms: interventions — PF-06372865; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1: (Experimental): Single ascending doses of PF-06372865 or placebo to investigate the safety/tolerability PK and PD of PF-06372865.
  Interventions: Drug: PF-06372865 or Placebo
- Cohort 2: (Experimental): Single ascending doses of PF-06372865 or placebo to investigate the safety/tolerability PK and PD of PF-06372865.
  Interventions: Drug: PF-06372865 or Placebo
- Cohort 3: (Experimental): Single ascending doses of PF-06372865 or placebo to investigate the safety/tolerability PK and PD of PF-06372865.
  Interventions: Drug: PF-06372865 or Placebo
- Cohort 4 (optional cohort): (Experimental): Two single doses of PF-06372865 or placebo or lorazepam to further investigate the pharmacodynamics of PF-06372865.
  Interventions: Drug: PF-06372865 or Placebo or Lorazepam

INTERVENTIONS:
Drug: PF-06372865 or Placebo — PF-06372865 will be administered as an extemporaneously prepared solution for all doses unless the tablet formulation need to be evaluated. Correspondingly, placebo doses will be administered as solution or tablet.
  Arms: Cohort 1:
Drug: PF-06372865 or Placebo — PF-06372865 will be administered as an extemporaneously prepared solution for all doses unless the tablet formulation need to be evaluated. Correspondingly, placebo doses will be administered as solution or tablet.
  Arms: Cohort 2:
Drug: PF-06372865 or Placebo — PF-06372865 will be administered as an extemporaneously prepared solution for all doses unless the tablet formulation need to be evaluated. Correspondingly, placebo doses will be administered as solution or tablet.
  Arms: Cohort 3:
Drug: PF-06372865 or Placebo or Lorazepam — Lorazepam 2 mg dose, PF-06372865 Dose 1, PF-06372865 Dose 2, PF-06372865 Dose 1 and Dose 2 in combination with lorazepam, placebo administered as tablet formulation
  Arms: Cohort 4 (optional cohort):

SUMMARY:
The purpose of this study in healthy people is to evaluate safety, toleration and time course of plasma concentration of single oral doses of PF-06372865. The pharmacodynamic activity of PF-06372865 will also be assessed. The effect of food on PK and the PK of PF-06372865 administered as a tablet formulation may also be investigated. Pharmacodynamic interaction between PF-06372865 and lorazepam will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects or female subjects of non-child bearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (e.g., gastrectomy).
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-dose
Apparent Oral Clearance (CL/F) | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-dose
Apparent Volume of Distribution (Vz/F) | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-dose
Plasma Decay Half-Life (t1/2) | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-dose
Area Under the Curve From Time Zero to 24 hours | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-dose
Change in Saccadic Eye Movements (saccadic reaction time, saccadic peak velocity and saccadic inaccuracy) | 0, 0.5, 1, 1.5, 2, 4, 6, 12 hours post-dose
Change in Body Sway | 0, 0.5, 1, 1.5, 2, 4, 6, 12 hours post-dose
Change in Smooth Pursuit | 0, 0.5, 1, 1.5, 2, 4, 6, 12 hours post-dose
Change in Bond and Lader VAS | 0, 0.5, 1, 1.5, 2, 4, 6, 12 hours post-dose
Change in Adaptive Tracking | 0, 0.5, 1, 1.5, 2, 4, 6, 12 hours post-dose
Change in Visual Verbal Learning Test | 1 and 6 hours post dose
Change in Pharmaco-EEG | 0, 0.5, 1, 1.5, 2, 4, 6, 12 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Leiden, CL, Netherlands

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7431001&StudyName=A%20First%20In%20Human%20Study%20In%20Healthy%20People%20To%20Evaluate%20Safety%2C%20Toleration%2C%20Pharmacokinetics%20and%20Pharmacodynamics%20of%20Single%20Oral%20Doses%20